CLINICAL TRIAL: NCT00194831
Title: Volumetric Brain Analysis in the Premature Brain: Correlation With Future Development
Brief Title: Correlation of Volumetric Brain Analysis With Development at 18 Months
Status: Withdrawn | Type: Observational
Why Stopped: No data. Study never completed.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Jeffrey Perlman, Weill Cornell
Other Study IDs: 000501007693
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
The study will correlate the volumes of the brain obtained from magnetic resonance imaging (MRI) scans done at term gestation for infants born prematurely who weighed less than 1000 grams at birth with their corresponding development at 18 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* All premature infants born < 1000 grams who had MRI scans of the brain at term gestation

Exclusion Criteria:

* Any known genetic or chromosomal abnormalities

Ages: 18 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants < 1000 gram birthweight who are followed post discharge as part of standard clinical care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Perlman, MB, Study Chair — New York Presbyterian Hospital Weill Cornell
Locations (1):
- New York Presbyterian Hospital Weill Cornell, New York, New York, United States